CLINICAL TRIAL: NCT02211950
Title: Evaluation of Relative Bioavailability of BI 44847 in Different Ethnic Groups (Subjects of White, Asian, and African Origin), and Evaluation of Effect of Diet and Acarbose Coadministration on Bioavailability Following Oral Administration of 200 mg BI 44847 in Healthy Male Volunteers. An Open-label, Single-dose, Parallel Group, Phase 1 Study (Group 1 With Additional Crossover Aspects)
Brief Title: Relative Bioavailability of BI 44847 in Different Ethnic Groups and Evaluation of Effect of Diet and Acarbose Coadministration on Bioavailability Following Oral Administration of 200 mg BI 44847 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1224.22
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Acarbose

ARMS (5):
- Treatment A (Experimental): single dose BI 44847 administered to white subjects
  Interventions: Drug: BI 44847
- Treatment B (Experimental): 100 mg acarbose for 2 days, on the second day a single dose BI 44847 administered to white subjects
  Interventions: Drug: BI 44847; Drug: Acarbose
- Treatment C (Experimental): single dose BI 44847 after a Japanese diet of 6 days administered to white subjects
  Interventions: Drug: BI 44847; Other: Japanese diet
- Treatment D (Experimental): single dose BI 44847 administered to asian subjects
  Interventions: Drug: BI 44847
- Treatment E (Experimental): single dose BI 44847 administered to african subjects
  Interventions: Drug: BI 44847

INTERVENTIONS:
Drug: BI 44847
Drug: Acarbose
  Other Names: Glucobay
  Arms: Treatment B
Other: Japanese diet
  Arms: Treatment C

SUMMARY:
The objectives were to investigate the relative bioavailability of BI 44847 in different racial groups (white, Asian, and African subjects) and to investigate the effect of different types of diet and acarbose coadministration on the bioavailability of BI 44847 in white subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects determined by results of screening
* Age 18 - 40 years
* Body Mass Index 18 - 25 kg/m2, at least 45 kg
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders as judged by the investigator
* Relevant gastrointestinal tract surgery
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or relevant neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts; systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, pulse rate out of 45 to 90 beats per minute
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use within 10 days prior to administration or during the trial of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation
* Participation in another trial with an investigational drug within 2 months after a multiple dose study or within 1 month after a single dose study
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 60 g/day in males, more than 40 g/day in females)
* Drug abuse, in the investigator's judgment upon review of the patient's history and urine screening for abused substances
* Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within 48 hours prior to trial or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance according to the assessment of the investigator
* Inability to comply with dietary regimen of study centre
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of the analyte in plasma in plasma over the time interval from 0 to infinity) | up to 48 hours after drug administration
AUC0-48 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 48 h) | up to 48 hours after drug administration
AUC0-12 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 12 h) | up to 48 hours after drug administration
Cmax (maximum concentration of the analyte in plasma) | up to 48 hours after drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
λz (terminal rate constant in plasma after single dose | up to 48 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma after single dose) | up to 48 hours after drug administration
MRTpo (mean residence time of the analyte in the body after single dose) | up to 48 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration after single dose) | up to 48 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz after single dose following extravascular administration) | up to 48 hours after drug administration
AUCt1-t2 (area under the concentration time curve of analyte in plasma over the time interval t1 to t2) | up to 24 hours after drug administration
Aet1-t2 (amount of drug that is eliminated in urine from the time point t1 to time point t2) | up to 24 hours after drug administration
fet1-t2 (fraction of drug eliminated in urine from time point t1 to time point t2) | up to 24 hours after drug administration
CLR,t1-t2 (renal clearance of the drug from the time point t1 until the time point t2) | up to 24 hours after drug administration
Amount of glucose excreted in urine | up to 24 hours after drug administration
Number of patients with adverse events | up to 48 hours after last administration of study drug
Number of patients with clinically relevant changes in laboratory tests | up to 48 hours after last administration of study drug
Number of patients with clinically relevant changes in Electrocardiogram (ECG) | up to 48 hours after last administration of study drug
Number of patients with clinically relevant changes in vital signs | up to 48 hours after last administration of study drug
Assessment of global tolerability by investigator on a 4-point scale | 48 hours after last administration of study drug